CLINICAL TRIAL: NCT00840502
Title: Impact of Malaria Infection in Pregnancy on Fetal and Newborn Growth
Brief Title: Ultrasound Study in Pregnant Women With Malaria
Acronym: UPS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU0801
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Pregnant Women; Malaria
Keywords: malaria; ultrasound; pregnancy; Pregnant women (infected with malaria and without)
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who present at the SMRU antenatal clinics on the Thai Burmese border.

SUMMARY:
Most of the neonatal deaths that occur worldwide every year are associated with low birth weight (LBW), caused by intrauterine growth restriction (IUGR) and/or preterm delivery. Accurate assessment of fetal growth and gestational age for timely identification and management of growth restriction are therefore public health priorities, especially in developing countries where 98% of all neonatal deaths occur. Every year, more than 50 million women become pregnant in malaria endemic regions. Malaria infection at any time during pregnancy reduces birthweight. However, little is known about the relationship between the timing of infection during pregnancy and the extent of the impact on birth weight. The mechanisms by which malaria causes LBW also remain unclear. Reduced placental blood flow, placental changes, red blood cell changes, severe anaemia and pro-inflammatory cytokines have all been implicated.

In this proposed, longitudinal, observational, minimal risk study, which will take place in SMRU antenatal clinics on the Thai-Burmese border, the effect of malaria infection during pregnancy on fetal growth will be determined. Women will be screened before 13+6 weeks of gestation and followed with regular ultrasound examinations during pregnancy. When a woman has a malaria infection an extra ultrasound scan will be done to measure growth retardation or placental blood flow changes. Bloodsamples will be taken to detect changes in red blood cell properties and putative markers of malaria infection. For this study the maximum amount of blood taken during pregnancy is 13 cc in an uninfected woman. For each malaria episode an additional 7 cc blood will be taken. After delivery a placenta and a cord sample will be taken to detect placental changes. The investigators aim to recruit four hundred pregnant women over the course of two years. This study involves minimal risk to participants as ultrasound examination is part of routine antenatal care in many countries in the world.

ELIGIBILITY:
Inclusion Criteria:

* Singleton viable pregnancy. If not detected at enrolment, multiple pregnancies will be excluded from the analysis.
* Age ≥18 years old.
* Willing and able to participate and comply with the study protocol and attend the SMRU ANCs regularly.
* EGA between 9+0 and 13+6 weeks by Ultrasound (CRL)
* Able to communicate in Burmese, Karen or English language
* written informed consent to participate in trial and follow consultation

Exclusion Criteria:

* Evidence of major congenital abnormality in the present pregnancy (e.g. anencephaly, omphalocele, hydrocephalus).
* Known chronic maternal illness.
* Thai national whose primary language is Thai

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregant women who present at the SMRU ante natal clinics. The antenatal clinics (ANC) are based on the Thai-Burmese border, in a region where Karen people (a minority group in Burma) are the principal inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 1887 (Actual)
Dates: Start 2009-02-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Ultrasound measurements | Up to birth

SECONDARY OUTCOMES:
Examination of all newborns | 6 months post natal

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Hashmi A, Carrara VI, Nyein PB, Darakamon MC, Charunwatthana P, McGready R. The Healthy Baby Flipbook: piloting home-based counseling for refugee mothers to improve infant feeding and water, sanitation, and hygiene (WASH) practices. Glob Health Action. 2019;12(1):1560115. doi: 10.1080/16549716.2018.1560115. PMID 31154995